CLINICAL TRIAL: NCT05332964
Title: Application of a Virtual Reliability System in the Evaluation of the Visual Spatial Attention in Stroke Patients
Brief Title: Virtual Reliability System for Visual Spatial Attention Evaluation in Stroke Patients
Status: Withdrawn | Type: Observational
Why Stopped: lack of time
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202104030RINC
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-02

CONDITIONS: Stroke Sequelae; Neglect, Hemispatial
Keywords: attention; hemineglect; virtual reality; reaction time
MeSH Terms: conditions — Perceptual Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- stroke (right): stroke patient with lesions at right hemisphere
- stroke (left): stroke patient with lesions at left hemisphere
- control: age-matched group for the stroke patients

SUMMARY:
The researchers designed a software based on a head-mounted displays for virtual reality (HMD-VR) to evaluate the reaction time to stimuli presented at right or left visual field. The study will recruit 100 stroke patients with hemisphere lesions (50 patients for right and left each) and 100 age-matched healthy controls. The participants will conduct a simple reaction time task in VR, with stimuli designated in the left or right hemi-field. The stroke patients will also received traditional tests for hemi-neglect. Test-retest reliability of the assessment will be conducted in a subset of the control group. The stroke patients will be followed in 3-4 weeks.

DETAILED DESCRIPTION:
The researchers designed a software based on a head-mounted displays for virtual reality (HMD-VR) to evaluate the reaction time to stimuli presented at right or left visual field. The study will recruit 100 stroke patients with hemisphere lesions (50 patients for right and left hemisphere each) and 100 age-matched healthy controls. The participants will conduct a simple reaction time task in VR, with stimuli designated in the left or right hemi-field. The stroke patients will also receive traditional tests for hemi-neglect. The researchers will also collect the demographic data, cognition function and daily activity function. Test-retest reliability of the assessment will be conducted in a subset of the control group. The stroke patients will be followed in 3-4 weeks. The researchers will compare the results of a traditional hemi-neglect tests and VR-based tests and their changes in two occasions.

ELIGIBILITY:
Inclusion Criteria for stroke patients:

1. aged at least 20 years old
2. diagnosed with stroke involving unilateral MCA and ACA territory
3. with unilateral upper limb with normal function
4. neurologically and medically stable.

Inclusion criteria for control group:

1) healthy adults, age-matched to stroke patients

Exclusion Criteria for both groups:

1. with history of neurological or psychiatric conditions other than stroke;
2. significant cognitive or speech problems that cause difficulties to cooperate with testing;
3. significant visual problems (such as color blindness, visual loss, cataract, glaucoma or other major eye condition)
4. upper limb musculoskeletal disorders to cause difficulties to use the keyboard or controller;
5. history of seizure, vestibular dysfunction or vertigo
6. can't tolerate HMD-VR

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: outpatient and inpatient rehabilitation unit in a medical center
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
reaction time | 4 weeks
  reaction time to the stimuli presented in the right or left hemi-field with VR software
hemineglect tests | 4 weeks
  Paper-based behavior inattention test (BIT)

SECONDARY OUTCOMES:
ADL | 4 weeks
  activities of daily living function evaluated by barthel index
cognition | 4 weeks
  using Montreal Cognitive Assessment (MoCA)
cybersickness | 1 day
  using Simulator Sickness Questionnaire (SSQ)

CONTACTS AND LOCATIONS:
Overall Officials: Huey-Wen Liang, MD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan